CLINICAL TRIAL: NCT00290537
Title: A Phase II Study of ZD6474 Alone and With Chemotherapy in Advanced NSCLC
Brief Title: Phase II Study of ZD6474 in Advanced NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual was suboptimal and increasing the number of patients was not feasible.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0635
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Carboplatin; Paclitaxel; ZD6474; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part One: ZD6474 (Experimental): First part of two part treatment, Part One: three 3-week cycles 300 mg of ZD6474 daily. Second part, Part Two: participants randomized to receive 300 mg of ZD6474 daily, or 100 mg of ZD6474 daily plus carboplatin AUC 6.0 intravenous (IV) over 15-30 minutes and paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 every 3 weeks.
  Interventions: Drug: ZD6474
- Part Two A: ZD6474 300 mg (Experimental): Second part of study where participants randomized to receive 300 mg of ZD6474 daily (group A)
  Interventions: Drug: ZD6474
- Part Two B: ZD6474 100 mg + Carboplatin + Paclitaxel (Experimental): Second part of study where participants randomized to receive 100 mg of ZD6474 daily plus carboplatin AUC 6.0 IV over 15-30 minutes and paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 every 3 weeks (group B).
  Interventions: Drug: ZD6474; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: ZD6474 — ZD6474 alone: Cycles 1-3 = 300 mg PO Daily x 3 Weeks; ZD6474+Carboplatin+Paclitaxel = 300 mg oral (PO) Daily or 100 mg PO Daily plus Carboplatin and Paclitaxel Every 3 Weeks.
  Other Names: Zactima; Vandetanib
Drug: Carboplatin — 6 AUC IV Over 15-30 Minutes, Immediately After Paclitaxel
  Other Names: Paraplatin
  Arms: Part Two B: ZD6474 100 mg + Carboplatin + Paclitaxel
Drug: Paclitaxel — 200 mg/m^2 IV Over 3 Hours On Day 1
  Other Names: Taxol
  Arms: Part Two B: ZD6474 100 mg + Carboplatin + Paclitaxel

SUMMARY:
The goal of this clinical research study is to learn how the drug ZD6474 affects the amount of tumor cell death in the body and the amount of blood that can be supplied to the tumor. The safety of ZD6474 alone and when given with chemotherapy will be studied. In addition, the side effects and response to this treatment will also be studied.

DETAILED DESCRIPTION:
ZD6474 is a new investigational drug that is thought to block the formation of new blood vessels. The growth of new blood vessels is called angiogenesis. Angiogenesis is thought to be essential for the growth of tumors beyond a small size. It is hoped that ZD6474 will limit new blood vessel growth in the tumor and "starve" the tumor by limiting blood flow to it. The second part of this study also includes paclitaxel (Taxol) and carboplatin (Paraplatin). Both paclitaxel and carboplatin are standard chemotherapy drugs that are approved by the FDA for use in the treatment of lung cancer.

Before beginning treatment on this study, you will have a biopsy of your tumor. The tissue taken during this biopsy will be compared with the tissue taken after you receive ZD6474. The tumor samples will be compared to see what effect ZD6474 has had on tumor cell death. During the biopsy procedure, you will receive either a local or general anesthetic depending on the location of your tumor and a small piece of tumor will be removed with a large needle.

Before treatment starts, you will have a complete physical exam by a physician. You will have routine blood (about 4 teaspoons) and urine tests. Women who are able to have children must have a negative blood pregnancy test. You will have a chest x-ray and a CT or MRI scan, a functional MRI, a bone scan if your doctor thinks it is necessary, and a brain scan. You will also have an ECG (test to measure the electrical activity of the heart) and a ECHO scan to make sure your heart is healthy enough to receive this treatment.

Treatment on this study will be given in 3-week cycles. During the first three cycles (i.e., the first 9 weeks) you will take a ZD6474 tablet by mouth each morning on an empty stomach. While on this study you will receive a physical exam every week. You will also receive weekly blood tests (about 4 teaspoons) for the first 4 weeks of treatment. After that you will receive blood tests (about 4 teaspoons) before every 3-week cycle.

After 2 weeks of treatment you will have another biopsy of your tumor, and another functional MRI. After every 9 weeks of treatment and every 2 cycles thereafter you will have a repeat CT or MRI to evaluate your tumor. If your disease has responded to ZD6474 or stayed the same, you will go on to the second part of this study. If your disease has gotten worse or intolerable side effects occur, you will be taken off this study and your doctor will discuss treatment options with you.

If you continue on to the second part of this study, you will be randomly assigned (as in the toss of a coin) to receive either: a) daily ZD6474 alone, or b) paclitaxel and carboplatin every 3 weeks along with daily ZD6474. You have an equal chance of being assigned to either group. If you receive paclitaxel, you will receive it as a 3-hour infusion into a vein on the first day of each treatment cycle. If you receive carboplatin, you will receive it by vein immediately following the paclitaxel infusion. The carboplatin infusion will take between 15 and 30 minutes. Treatment with either daily ZD6474 or ZD6474 plus paclitaxel and carboplatin will continue until your diseases worsens or until severe side effects occur.

This is an investigational study. ZD6474 is an investigational drug that has been approved by the FDA for research use only. A total of up to 120 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent form must be completed before any protocol specific screening. Patient must consent to a tissue biopsy at study entry and again at the week 3.
2. Patients must have a diagnosis of stage IIIb or stage IV non-small cell lung cancer (histologically or cytologically proven) and must not be eligible for combined chemotherapy and radiation therapy.
3. Patients must have at least one site of measureable disease that is amenable to biopsy. The patient must not have had radiation to this site. Lesion must be at least 20 mm in the longest diameter by spiral CT or 20 mm with conventional techniques according to RECIST.
4. Eligible patients must have an ECOG performance status of 0-1.
5. Patients must have adequate hepatic, renal, and bone marrow function as defined below: 1) Serum creatinine < 1.5 mg/dL or a calculated creatinine clearance > 60 mL/min 2)· Total bilirubin < 1.5 x ULN ·3) ALT or AST </= 2.5 x ULN OR ALT or AST </= 5.0 x ULN if related to liver metastases OR Alk Phos </= 2.5 x ULN ·4) WBC > 3,000/mm**3 ·5) ANC > 1,500 mm**3 ·6) Platelets > 100,000/mm**3 ·7) Hemoglobin > 10 g/dL ·8) PT/PTT < 1.5 x normal
6. Patients must be >= 18 years of age.

Exclusion Criteria:

1. Patients are excluded if they have received prior chemotherapy for this disease type.
2. Patients with brain metastases are not eligible for this study unless treated at least 4 weeks before entry and stable without steroid treatment for 1 week.
3. Prior radiation therapy allowed to <25% of the bone marrow. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.
4. Patients may not have any concomitant uncontrolled medical or psychiatric disorders.
5. Patients must not be pregnant or breast-feeding. All women of childbearing potential must have a negative pregnancy test. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy. There is no specific information available on the effects of this drug on women who are pregnant or breast-feeding. Therefore these patients are excluded from this study because of the unknown risks involved. All sexually active patients must practice adequate contraception for the entire treatment period.
6. Patients must not have undergone minor surgery (e.g., central venous catheter placement) within 24 hours of treatment with ZD6474. Patients may not have undergone any major surgery (e.g., laparotomy, thoracotomy, or craniotomy) within four weeks of enrollment.
7. Patients may not have a history of a bleeding diathesis.
8. Patients must agree not to use herbal remedies or other over-the-counter biologics (e.g., shark cartilage)
9. Significant cardiac event (including symptomatic heart failure or angina) within 3 months of entry or presence of cardiac disease that in the opinion of the Investigator increase the risk of ventricular arrythmia.
10. History of clinically significant arrhythmia (multifocal PVCs, bigeminy, trigeminy, ventricular tachycardia) which is symptomatic or requires treatment (CTC grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
11. Presence of left bundle branch block (LBBB).
12. Previous history of QT prolongation as a result from other medication that required discontinuation of that medication.
13. Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
14. QTc with Bazett's correction that is unmeasurable, or >/= 480 msec on screening ECG. If a patient has QTc >/= 480 msec on screening ECG, the screening may be repeated twice (at least 24 hours apart). The average QTc from the 3 screening ECGs must be < 480 msec in order for the patient to be eligible for the study.
15. Any concomitant medications that may cause QTc prolongation or induce Torsades de Pointes (see Appendix F) or induce CYP3A4 function (see section 8.2).
16. Potassium level less than 3.5 meq/l; calcium and magnesium level outside normal limits. Supplementation of electrolytes is permitted.
17. Left ventricular ejection fraction less than 45% measured by echocardiogram for subjects with previous anthracycline therapy (total dose greater than 450 mg/m2), significant cardiovascular disease, or chest irradiation
18. History of severe hypersensitivity reaction to drugs formulated with polysorbate 80
19. Any concurrent condition which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
20. Participation in an investigational trial within the past 30 days.
21. Because of DCE-MRI, individuals with the following are excluded: 1) Cardiac pacemakers or neurostimulators, 2) Metal implants other than those approved as being safe in an MRI environment, 3) Claustrophobia, 4) Physical characteristics that preclude a MRI scan
22. Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
23. Currently active diarrhea that may affect the ability of the patient to absorb the ZD6474 or tolerate diarrhea.
24. Previous or current malignancies at other sites within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell carcinoma or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D.Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/19/2006 through 11/03/2006. All participants recruited at University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Part Two: ZD6474 + Carboplatin + Paclitaxel: Second part of two part treatment, Part One /Two: participants randomized to receive 300 mg of ZD6474 daily, or 100 mg of ZD6474 daily plus carboplatin AUC 6.0 intravenous (IV) over 15-30 minutes and paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 every 3 weeks.
Period: Overall Study
Arm/Group | Part One: ZD6474 | Part Two: ZD6474 + Carboplatin + Paclitaxel
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ZD6474: Part One: three 3-week cycles 300 mg of ZD6474 daily.
Arm/Group | ZD6474
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 50 [35 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Following Treatment With 300 mg ZD6474 Daily (Study Part One)
Description: Evaluate the response rate in patients receiving monotherapy with ZD6474 compared to ZD6474 plus carboplatin plus paclitaxel. No formal comparisons could be made and no conclusions drawn because of small numbers in the treatment groups; a result of an inability to fulfil the recruitment target.
Time Frame: Radiologic evaluations performed after weeks 2 and 9 of treatment, then every 2 cycles or as indicated if progressive disease is suspected up to 6 cycles or 18 weeks (1 cycle = 3 weeks).
Measure: Number; unit: Participants
Groups:
- ZD6474: First part of treatment: three 3-week cycles 300 mg of ZD6474 daily. Second part, patients randomized to receive 300 mg of ZD6474 daily, or 100 mg of ZD6474 daily plus carboplatin and paclitaxel every 3 weeks.
- ZD6474 + Carboplatin + Paclitaxel: Second part, patients randomized to receive 300 mg of ZD6474 daily, or 100 mg of ZD6474 daily plus carboplatin and paclitaxel every 3 weeks.
Arm/Group | ZD6474 | ZD6474 + Carboplatin + Paclitaxel
Number analyzed (Participants) | 4 | 0
Participants
  Complete Response | 1 |
  No Change/Stable Disease | 1 |
  Progressive Disease | 1 |
  Inevaluable for Response | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events collected through three 3-week cycles, then up to two weeks after treatment.
Arm/Group | ZD6474
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD6474 (N=4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
Alanine aminotransferase increased (ALT, SGPT) (Investigations) | 2 (2)
ANOREXIA (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (AST, SGOT) (Investigations) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EDEMA: LIMB (General disorders) | 1 (1)
ERYTHEMA MULTIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
FATIGUE (General disorders) | 2 (2)
HEMOGLOBIN INCREASED (Investigations) | 1 (1)
HEMORRHAGE, PULMON (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHAGE/BLEEDIN (Blood and lymphatic system disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
INCONTINENCE, ANAL (Gastrointestinal disorders) | 1 (1)
LYMPHOPENIA (Vascular disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
NAUSEA ALONE (Gastrointestinal disorders) | 1 (1)
VISION LOW (Eye disorders) | 2 (2)
PAIN (ABDOMEN NOS) (Gastrointestinal disorders) | 1 (1)
PAIN (EYE) (Eye disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No